CLINICAL TRIAL: NCT05454202
Title: Assessment of the Interest of ANI in the Non-communicating Patient in Palliative Care
Acronym: ANI-CARE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0830; 2022-A00631-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: End of Life; Pain; Analgesia
Keywords: Analgesia/Nociception Index; end-of-life, comfort evaluation, comfort monitoring, palliative care, non-communicating; comfort evaluation; comfort monitoring; palliative care; non-communicating
MeSH Terms: conditions — Death; Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-communicating: Non-communicating (Glasgow ≤ 10) end-of-life patient hospitalized in palliative care (age ≥ 18 years old)
  Interventions: Device: ANI

INTERVENTIONS:
Device: ANI — Pain measurement during care procedures in palliative care

SUMMARY:
Comfort evaluation is one of the major challenges in the palliative care setting, particularly when it comes to non-communicative patients. ANI monitoring is a non-invasive and painless technique which evaluates the parasympathetic tone activity through heart rate variability. It has proven reliable for pain assessment during general anesthesia (GA) or for sedated critically ill patients. The parasympathetic activity seems to be a good reflect of the patient's comfort, implicating stress and anxiety.

So, the ANI could be an interesting tool to assess the comfort of non-communicating end-of-life patients.

That is why the goal of our study is to assess the interest of ANI to assess the comfort of non-communicating patients hospitalized in palliative care during a painful care by comparing the ANI measure to the CPOT scale realised by the nurses in a blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in palliative care Non-communicating patients (Glasgow ≤ 10)

Exclusion Criteria:

* Non sinusal heart rate
* Respiratory rate < 9/min
* Treated by inotropes
* Pace-maker
* Patient in agonal phase
* Opposition from the guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-communicating end-of-life patient hospitalized in palliative care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Variation of the ANI between before the care and during the care | From 10 minutes before the care to 10 minutes after the care

SECONDARY OUTCOMES:
Variation of the ANI between during the care and after the care | From 10 minutes before the care to 10 minutes after the care
Coefficient of correlation between the variation of the ANI and the variation of the CPOT scale between each periods. | From 10 minutes before the care to 10 minutes after the care
Coefficient of correlation between the minANI and the CPOT scale for each periods | From 10 minutes before the care to 10 minutes after the care
Coefficient of correlations between ANImin and CPOT values before, during, and after the painful care session | From 10 minutes before the care to 10 minutes after the care
The discriminatory power of the ANI to separate the non-comfortable and the comfortable population defined by a ≤ 2 threshold on the CPOT scale | From 10 minutes before the care to 10 minutes after the care

CONTACTS AND LOCATIONS:
Overall Officials: Chloe PRODHOMME, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Cardiologique Chu Lille, Lille, France